CLINICAL TRIAL: NCT00645632
Title: Treatment of Newly Diagnosed Untreated Osteosarcoma: A Pilot Study of a New Chemotherapeutic Regimen Including Ifosfamide
Brief Title: Combination Chemotherapy in Treating Patients Undergoing Surgery for Newly Diagnosed High-Grade Osteosarcoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Carola A.S. Arndt, Mayo Clinic
Purpose: Treatment
Other Study IDs: CDR0000582263; P30CA015083 (NIH); 909101 (Other: Mayo Clinic Cancer Center); 549-90 (Other: Mayo Clinic IRB)
Record Dates: First submitted 2008-03-26; First posted 2008-03-27 (Estimated); Last update posted 2011-05-16 (Estimated); Status verified 2011-05

CONDITIONS: Sarcoma
Keywords: localized osteosarcoma
MeSH Terms: conditions — Sarcoma | interventions — Cisplatin; Doxorubicin; Ifosfamide; Methotrexate; Chemotherapy, Adjuvant; Neoadjuvant Therapy

INTERVENTIONS:
Drug: cisplatin
Drug: doxorubicin hydrochloride
Drug: ifosfamide
Drug: methotrexate
Procedure: adjuvant therapy
Procedure: neoadjuvant therapy
Procedure: therapeutic conventional surgery

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as ifosfamide, methotrexate, cisplatin, and doxorubicin, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving chemotherapy before surgery may make the tumor smaller and reduce the amount of normal tissue that needs to be removed. Giving it after surgery may kill any tumor cells that remain after surgery.

PURPOSE: This clinical trial is studying how well combination chemotherapy works in treating patients undergoing surgery for newly diagnosed high-grade osteosarcoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* To evaluate the efficacy of a new induction regimen comprising ifosfamide in combination with high-dose methotrexate, cisplatin, and doxorubicin hydrochloride, in terms of clinical response and pathological response of the tumor, in patients with newly diagnosed high-grade osteosarcoma.
* To determine the overall survival and disease-free survival of these patients.
* To evaluate the toxicity of this regimen.
* To correlate MRI imaging of the primary tumor with histopathologic grading after treatment with this regimen.

OUTLINE: This is a multicenter study.

* Neoadjuvant chemotherapy (weeks 1-15): Patients receive ifosfamide IV over 1 hour on days 1-5 and 36-40; doxorubicin hydrochloride IV over 18 hours on days 1-3 and 36-38 and IV over 72 hours on days 71-73; high-dose methotrexate IV over 4 hours on days 22, 29, 57, 64, 92, and 99; and cisplatin IV over 4 hours on day 71.
* Surgery (week 16): Patients undergo resection of the tumor on day 106. Patients found to have unresectable disease are treated on an alternative protocol unless they have clear clinical and pathologic response to treatment.
* Adjuvant chemotherapy (weeks 18-43): Beginning 2 weeks after surgery, patients receive ifosfamide IV over 1 hour on days 120-124, 155-159, 225-229, and 260-264; doxorubicin hydrochloride IV over 18 hours on days 120-122 and 155-157 and IV over 72 hours on days 190-192; high-dose methotrexate IV over 4 hours on days 141, 148, 176, 183, 211, 218, 246, 253, 281, and 288; and cisplatin IV over 4 hours on days 190 and 289.

After completion of study therapy, patients are followed every 2 months for 1 year, every 4 months for 2 years, every 6 months for 2 years, and then annually thereafter.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed osteosarcoma of the extremity

  * High-grade (grade III or IV) disease

    * No low-grade disease (e.g., parosteal or periosteal osteosarcoma)
* No secondary osteosarcoma (i.e., tumor occurring in a radiotherapy field designed for a prior tumor)
* No Paget's disease
* No known metastases

PATIENT CHARACTERISTICS:

* Total bilirubin < 2 times normal
* AST < 2 times normal
* Alkaline phosphatase < 2 times normal
* Creatinine ≤ 1.5 mg/dL OR creatinine clearance > 60 mL/min
* LVEF ≥ 45%
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No other prior malignancy except retinoblastoma

  * Patients with familial retinoblastoma syndrome who develop osteosarcoma unrelated to radiotherapy (e.g., in a primary site in the extremities) are eligible

PRIOR CONCURRENT THERAPY:

* No prior chemotherapy or radiotherapy

  * Patients with retinoblastoma may have received radiotherapy to the orbits
* At least 28 days since prior initial amputation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 1990-11; Primary Completion 1995-01 (Actual); Study Completion 2008-01 (Actual)

PRIMARY OUTCOMES:
Histopathologic response rate
Clinical response rate
Toxicity
Disease-free survival
Overall survival

CONTACTS AND LOCATIONS:
Overall Officials: Gerald S. Gilchrist, MD, Study Chair — Mayo Clinic; Tom R Fitch, M.D., Principal Investigator — Mayo Clinic; Gerardo Colon-Otero, M.D., Principal Investigator — Mayo Clinic